CLINICAL TRIAL: NCT03787303
Title: A Single Arm Phase II Pilot Study of Euthyroid Hypothyroxinemia in Metastatic Breast Carcinoma
Brief Title: Study of Euthyroid Hypothyroxinemia in Metastatic Breast Carcinoma
Acronym: B-TREUH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Relocation of Principal Investigator
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Principal Investigator, Shruti Trehan MD, Shruti Trehan MD, Aultman Health Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.08.ST
Record Dates: First submitted 2018-12-12; First posted 2018-12-26 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Breast Cancer; Thyroid Dysfunction
MeSH Terms: conditions — Breast Neoplasms | interventions — Triiodothyronine

STUDY DESIGN:
Intervention Model Description: Triiodothyronine (T3) - IND Exempt
Masking Description: N/A (not applicable)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Triiodothyronine (T3) (Experimental): Following discontinuation of L-thyroxine (T4), triiodothyronine (T3) will be initiated at a 3:1 ratio. The dose will be titrated by the investigator to maintain levels of free T4 < 50% of normal range while maintaining a euthyroid state. Triiodothyronine (T3) tablets for oral administration will be prescribed once or twice daily depending on the total dose. Treatment duration will be approximately 9 months during which time the subjects will continue to be treated and monitored as usual for their metastatic breast cancer. During the study period and at the conclusion of the study period, there will be continuous evaluations of the disease status and thyroid status with the option of resuming the original thyroid replacement or continuation of the triiodothyronine (T3).
  Interventions: Drug: Triiodothyronine (T3)

INTERVENTIONS:
Drug: Triiodothyronine (T3) — Participants will have their L-thyroxine (T4) discontinued and Triiodothyronine (T3)/liothyronine sodium initiated at 3: 1 and titrated.
  Other Names: liothyronine sodium

SUMMARY:
Up to one third of breast cancer patients have hypothyroidism or hyperthyroidism. L-thyroxine (T4), or Synthroid, is the most commonly prescribed agent for the management of hypothyroidism in the US. However, there are data suggesting that triiodothyronine (T3) may have benefits in preventing disease progression over l-thyroxine (T4).

DETAILED DESCRIPTION:
It is estimated that there are approximately 155,000 living with metastatic breast cancer in the US and the number is estimated to increase over the next years (SEER data). Although their median survival has improved over the last 2 decades from 17 months to approximately 24 months attributed to newer treatments, there is an ongoing need for additional strategies and research to improve survival and quality of life.

Many studies have explored the connection between hypothyroidism and hyperthyroidism and breast cancer with varied results ranging up to one third prevalence. Low Triiodothyronine (T3) and elevated Thyroid-Stimulating Hormone (TSH) levels have been detected in newly diagnosed breast cancer patients. Other studies have suggested that some of the common symptoms reported by breast cancer survivors such as fatigue and depression can be attributed to subclinical hypothyroidism.

L-thyroxine (T4) is the most commonly prescribed agent for the management of hypothyroidism in the US. However, there are data suggesting that T4 is a potent pro-oncogenic agent. Proposed mechanisms include stimulation of mitogenesis, angiogenesis and resistance to apoptosis, opposition of anti-PDL-1 and radiation effects. It has been postulated that the avbeta3integrin that is universally expressed on cancer cells harbors a thyroid hormone receptor and T4 interacts with it.

Triiodothyronine (T3) on the other hand, is significantly less oncogenic and less mitogenic and is downstream of T4 which is a T3 pro-hormone. Therefore, exogenous supplementation of T3 would decrease the T4 levels creating the desired state of euthyroid hypothyroxinemia.

The rationale of this study is to replace L-thyroxine (T4) with Triiodothyronine (T3) in hypothyroid patients with metastatic breast carcinoma while they continue to receive standard systemic therapy, titrating the dose to achieve a state of euthyroid hypothyroxinemia which is turn would result in a lower risk of disease progression and improved survival by lowering the concentration of T4.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* Male or female with diagnosis of metastatic breast carcinoma and documented history of hypothyroidism .
* TSH level within normal range at baseline
* Life expectancy estimated > 3 months
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Life expectancy estimated to be less than 3 months
* Is currently pregnant or intends to become pregnant during the duration of the study
* Active angina, New York Heart Association (NYHA) advanced [Class III/IV] congestive heart failure, or uncontrolled cardiac arrhythmia within 6 months of enrollment
* History of thyrotoxicosis
* History of adrenal insufficiency
* Hypersensitivity to any active or extraneous constituents in Triiodothyronine (T3)/liothyronine sodium

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Trehan, MD, Principal Investigator — Aultman Health Foundation
Locations (1):
- Aultman Medical Group Hematology and Oncology, Canton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 participants from one local medical oncology practice were enrolled between March 1, 2019 and March 9, 2022.
Pre-assignment Details: All enrolled participants underwent a four day washout period of L-thyroxine (T4) prior to Triiodothyronine (T3) initiation. There were no enrolled participants who were excluded from the study.
Period: Overall Study
Arm/Group | Triiodothyronine (T3)
Started | 7
Completed | 5
Not Completed | 2
Not completed — Death | 1
Not completed — Premature Termination of Study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Triiodothyronine (T3)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
Duration of time since diagnosis of metastatic disease [Mean (Standard Deviation); unit: months] | 62.1 (79.52)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival at 12 Months Based Upon Clinical and Radiological Assessments Completed as Part of Routine Care
Description: To prospectively evaluate the progression-free survival in hypothyroid patients with metastatic breast carcinoma who are rendered euthyroid and hypothyroxinemic. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the nadir sum of the longest diameter (SLD) of target lesions, or unequivocal progression (overall level of substantial worsening) in existing non-target lesions, or the appearance of one or more new lesions.
Time Frame: 12 months
Population: Last enrolled subject was only able to be followed for 9 months due to early termination of study. Subject not included in primary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Triiodothyronine (T3)
Number analyzed (Participants) | 6
Participants | 4

2. Secondary Outcome: Number of Patients With Both Metastatic Breast Cancer and Hypothyroidism in All Screened Patients.
Description: To quantitate the prevalence of hypothyroidism in metastatic breast cancer patients at a community oncology practice.
Time Frame: Study duration, planned was 48 months but actual was 36 months [March 1, 2019 to March 9, 2022] due to premature closure due to planned relocation of the PI.
Population: Outcome was number of practice patients with both metastatic breast cancer and hypothyroidism. Of the 26 identified, 7 patients consented to enroll on the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Triiodothyronine (T3)
Number analyzed (Participants) | 126
Participants | 26

3. Secondary Outcome: Measurement of Quality of Life Total Score Across Time Using Validated FACT-B Questionnaire
Description: Functional Assessment of Cancer Therapy - Breast (FACT-B) Total Score comprised of Physical Well Being (PWB), Social Well Being (SWB), Emotional Well Being (EWB), Functional Well Being (FWB), and Breast Cancer Subscale (BCS). Range is 0-148. A higher score indicates higher quality of life. Missing scores were handled by prorating values.
Time Frame: Baseline, 3, 6, 9, and 12 months
Population: Of the 7 subjects enrolled only 5 of the patients completed Quality of Life FACT-B questionnaires for all five timepoint. Two subjects did not complete the 12 months surveys due to death or premature study termination.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triiodothyronine (T3)
Number analyzed (Participants) | 7
score on a scale
  Baseline | 114 (24.56)
  At 3 months | 114 (16.80)
  At 6 months | 116 (20.71)
  At 9 months | 112 (26.92)
  At 12 months: number analyzed (Participants) | 5
  At 12 months | 110 (23.68)

4. Secondary Outcome: Measurement of Energy Level Across Time Using FACT-B Question.
Description: Functional Assessment of Cancer Therapy - Breast (FACT-B) Lack of energy on 5 point Likert scale as measured on FACT-B Physical Well-being subscale. Score of 0 indicates no lack of energy with score of 4 indicating total lack of energy.
Time Frame: Baseline, 3, 6, 9, 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triiodothyronine (T3)
Number analyzed (Participants) | 7
score on a scale
  Baseline | 2.9 (1.07)
  3 months | 2.4 (1.3)
  6 months | 3.0 (1.16)
  9 months | 3.0 (1.53)
  12 months: number analyzed (Participants) | 5
  12 months | 2.6 (1.14)

5. Secondary Outcome: Time to Achieve Euthyroid Hypothyroxinemia State
Description: To study the average time required to achieve euthyroid hypothyroxinemia state in qualifying patients. Thyroid function laboratory testing was performed at baseline and then at every 4 weekly intervals until 12 weeks then every 3 monthly thereafter, unless thyroid-stimulating hormone (TSH) was abnormal. If a normal TSH level was not achieved by the 12 week visit, repeat TSH measurements were ordered every 4-6 weeks until the TSH value was within the laboratory normal reference range. Initial euthyroid state defined by number of days between initiation of triiodothyronine (T3) and documentation of first normal TSH value.
Time Frame: Number of days between initiation of triiodothyronine (T3) and documentation of first normal TSH value for each participant, assessed up to 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Triiodothyronine (T3)
Number analyzed (Participants) | 7
days | 59.6 (50.64)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each subject at every 3 monthly visit and is reported as below. Attribution or etiology under comments below. Study period was 12 months (9 months for last patient due to premature termination of study)
Description: 112/124 - 88.7% of adverse events were deemed to be related to underlying metastatic breast cancer and/or treatment thereof.
  0 events reported definitely related to the study drug 14/124 -11.3% events reported as possible or probably related to the study drug Cause of mortality reported due to metastatic breast cancer.
Arm/Group | Triiodothyronine (T3)
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triiodothyronine (T3) (N=7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
ascites (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triiodothyronine (T3) (N=7)
Edema limbs (General disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2)
Memory Impairment (Nervous system disorders) | 3 (3)
Hypertension (Vascular disorders) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bronchial infection (Infections and infestations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder: Other hemoccult positive (Gastrointestinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Skin disorder other: Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Endocrine disorder: Cold intolerance (Endocrine disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Weight loss (Investigations) | 2 (2)
Headache (Nervous system disorders) | 2 (4)
Chills (General disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Arthalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Gastrointestinal disorders: Other - Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Skin disorder: Other - Chest wall redness (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Anosmia (Nervous system disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder: Other-onycholysis (Skin and subcutaneous tissue disorders) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Alopecia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (4)
White blood cell count decreased (Investigations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4)
Blood bilirubin increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decrease (Investigations) | 3 (5)
Blood urea nitrogen increase (Renal and urinary disorders) | 1 (2)
Creatinine increase (Renal and urinary disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Nail peeling (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitation is small sample size due to pandemic affecting clinical trial accrual. A larger sample is needed to adequately answer the research question.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03787303/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT03787303/SAP_003.pdf
  • Informed Consent Form (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT03787303/ICF_002.pdf